CLINICAL TRIAL: NCT00343863
Title: Efficacy of Palonosetron in the Prevention of Acute and Delayed Chemotherapy-Induced Nausea and Vomiting Following Dose Dense Adriamycin-Cyclophosphamide Chemotherapy in Early Stage Breast Cancer Patients
Brief Title: Dexamethasone and Ondansetron Hydrochloride or Palonosetron Hydrochloride in Preventing Nausea and Vomiting in Patients Receiving Doxorubicin Hydrochloride and Cyclophosphamide For Early Stage Breast Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Hannah Linden, Principal Investigator, University of Washington
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Supportive Care
Other Study IDs: 6140; NCI-2010-00801 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2006-06-22; First posted 2006-06-23 (Estimated); Results first posted 2017-07-11 (Actual); Last update posted 2017-07-11 (Actual); Status verified 2017-06

CONDITIONS: Male Breast Cancer; Nausea and Vomiting; Stage I Breast Cancer; Stage II Breast Cancer; Stage IIIA Breast Cancer
MeSH Terms: conditions — Breast Neoplasms, Male; Nausea; Vomiting; Breast Neoplasms | interventions — Palonosetron; Cyclophosphamide; Dexamethasone; Calcium Dobesilate; Doxorubicin; Therapeutics; Ondansetron

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Dexamethasone + Ondansetron IV on Day 1 (Active Comparator): All patients receive doxorubicin hydrochloride IV on day 1 and oral cyclophosphamide on days 1-7.
  Patients receive dexamethasone IV or orally and ondansetron IV on day 1 (prior to each dose of doxorubicin hydrochloride).
  Interventions: Drug: cyclophosphamide; Drug: dexamethasone; Drug: doxorubicin hydrochloride; Procedure: quality-of-life assessment; Procedure: nausea and vomiting therapy; Procedure: management of therapy complications; Drug: ondansetron hydrochloride; Other: survey administration
- Dexamethasone + Palonosetron IV on Day 1 (Experimental): All patients receive doxorubicin hydrochloride IV on day 1 and oral cyclophosphamide on days 1-7.
  Patients receive dexamethasone IV or orally and palonosetron IV on day 1 (prior to each dose of doxorubicin hydrochloride).
  Interventions: Drug: palonosetron hydrochloride; Drug: cyclophosphamide; Drug: dexamethasone; Drug: doxorubicin hydrochloride; Procedure: quality-of-life assessment; Procedure: nausea and vomiting therapy; Procedure: management of therapy complications; Other: survey administration

INTERVENTIONS:
Drug: palonosetron hydrochloride — Given IV
  Other Names: Aloxi; RS 25259-197
  Arms: Dexamethasone + Palonosetron IV on Day 1
Drug: cyclophosphamide — Given orally
  Other Names: CPM; CTX; Cytoxan; Endoxan; Endoxana
Drug: dexamethasone — Given orally or IV
  Other Names: Aeroseb-Dex; Decaderm; Decadron; DM; DXM
Drug: doxorubicin hydrochloride — Given IV
  Other Names: ADM; ADR; Adria; Adriamycin PFS; Adriamycin RDF
Procedure: quality-of-life assessment — Ancillary studies
  Other Names: quality of life assessment
Procedure: nausea and vomiting therapy — Given IV
  Other Names: antiemetic support; management of nausea and vomiting; nausea and vomiting management; therapy, nausea and vomiting; vomiting and nausea management
Procedure: management of therapy complications — Given IV
  Other Names: complications of therapy, management of
Drug: ondansetron hydrochloride — Given IV
  Other Names: GR 38032F; GR-C507/75; SN-307; Zofran
  Arms: Dexamethasone + Ondansetron IV on Day 1
Other: survey administration — Ancillary studies

SUMMARY:
RATIONALE: Antiemetic drugs, such as dexamethasone, ondansetron hydrochloride, and palonosetron hydrochloride, may help lessen or prevent nausea and vomiting caused by chemotherapy.

PURPOSE: This clinical trial studies how well giving dexamethasone together with ondansetron hydrochloride or palonosetron hydrochloride works in preventing nausea and vomiting in patients receiving doxorubicin hydrochloride and cyclophosphamide for early stage breast cancer

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the proportion of patients achieving a complete response (CR), defined as no emesis and no rescue medications in the 0-24 hour time period following weekly intravenous doxorubicin.

SECONDARY OBJECTIVES:

I. To determine the proportion of patients achieving a complete response (CR), defined as no emesis and no rescue medications in the 24-120 hour time period following weekly intravenous doxorubicin.

II. To determine the proportion of patients achieving a complete response (CR), defined as no emesis and no rescue medications in the 0-120 hour time period following weekly intravenous doxorubicin.

III. To determine the number of emetic episodes daily and cumulatively for the 24-120, and 0-120 hour time periods.

IV. To determine the time to first emetic episode. V. To determine the time to first administration of rescue medication. VI. To determine the time to treatment failure (time to first emetic episode or administration of rescue medication, whichever occurred first).

VII. To determine the number of doses of rescue medications used. VIII. To determine the side effects of antiemetic medications used. IX. To determine theseverity of nausea. X. To evaluate quality of life.

OUTLINE: Patients are assigned to 1 of 2 treatment groups.

All patients receive doxorubicin hydrochloride IV on day 1 and oral cyclophosphamide on days 1-7.

GROUP I: Patients receive dexamethasone IV or orally and ondansetron IV on day 1 (prior to each dose of doxorubicin hydrochloride).

GROUP II: Patients receive dexamethasone IV or orally and palonosetron IV on day 1 (prior to each dose of doxorubicin hydrochloride).

Treatment repeats every 7 days for 12-15 courses in the absence of disease progression or unacceptable toxicity.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have a histologically confirmed diagnosis of primary breast carcinoma
* Patient must be naive to chemotherapy at the time of enrollment
* Patients must have prescribed weekly intravenous adriamycin (doxorubicin) and daily oral cyclophosphamide treatment for early breast cancer
* The patient must be informed of the investigational nature of this study and must sign and give written informed consent in accordance with institutional and federal guidelines
* Patients must have a Karnofsky index of greater than or equal to 50%
* Known mild to moderate hepatic, renal or cardiovascular impairment may be enrolled at the discretion of the investigator

Exclusion Criteria:

* Receipt of investigational drug within 30 days before study entry
* Received any drug with potential anti-emetic effect within 24 hours prior to the start of study-designated chemotherapeutic agent (with the exception of administration of the palonosetron/dexamethasone infusion solution), including the following: 5-HT3 receptor antagonists; dopamine receptor antagonists (metoclopramide); phenothiazine anti-emetics (prochlorperazine, thiethylperazine and perphenazine); diphenhydramine, scopolamine, chlorpheniramine maleate, trimethobenzamide (diphenhydramine will be allowed if given for prophylactic treatment of hypersensitivity reactions associated with the administration of Taxanes); all benzodiazepines; haloperidol, droperidol, tetrahydrocannabinol, or nabilone; any systemic corticosteroid (hydrocortisone, methylprednisolone, prednisone) (topical or inhaled preparations are allowed)
* Any vomiting, retching or NCI Common Toxicity Criteria version 3.0 grade 2-4 nausea in the 24 hours preceding chemotherapy
* Ongoing vomiting from any organic etiology
* Need to receive systemic corticosteroids, except: a) when defined as part of the chemotherapy regimen as a preventative measure for chemotherapy toxicities; b) topical or inhaled preparations; and/or c) when used as rescue medication during the study
* Known contraindication to 5-HT3 receptor antagonists (including palonosetron) or dexamethasone
* Need to receive radiotherapy during the study
* Inability to understand or cooperate with study procedures

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2006-01; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hannah Linden, Principal Investigator — Fred Hutchinson Cancer Research Center/University of Washington Cancer Consortium
Locations (1):
- Fred Hutchinson Cancer Research Center/University of Washington Cancer Consortium, Seattle, Washington, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Dexamethasone + Ondansetron IV: All patients receive doxorubicin hydrochloride IV on day 1 and oral cyclophosphamide on days 1-7.
  Patients receive dexamethasone IV or orally and ondansetron IV on day 1 (prior to each dose of doxorubicin hydrochloride).
- Dexamethasone + Palonosetron IV: All patients receive doxorubicin hydrochloride IV on day 1 and oral cyclophosphamide on days 1-7.
  Patients receive dexamethasone IV or orally and palonosetron IV on day 1 (prior to each dose of doxorubicin hydrochloride).
Period: Overall Study
Arm/Group | Dexamethasone + Ondansetron IV | Dexamethasone + Palonosetron IV
Started | 7 | 34
Completed | 7 | 34
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Dexamethasone + Ondansetron IV | Dexamethasone + Palonosetron IV | Total
Number analyzed (Participants) | 7 | 34 | 41
Age, Continuous [Median (Full Range); unit: years] | 54 [45 to 63] | 49 [29 to 69] | 50 [29 to 69]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 34 | 41
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 2 | 3
  Not Hispanic or Latino | 6 | 30 | 36
  Unknown or Not Reported | 0 | 2 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 6 | 31 | 37
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 2 | 2

OUTCOME MEASURES:

1. Primary Outcome: Count of Patients Achieving a Complete Response
Time Frame: At 0-24 hours after weekly intravenous doxorubin
Measure: Count of Participants; unit: Participants
Arm/Group | Dexamethasone + Ondansetron IV | Dexamethasone + Palonosetron IV
Number analyzed (Participants) | 7 | 34
Participants | 3 | 15

2. Secondary Outcome: Count of Patients Achieving Complete Response
Time Frame: At 24-120 hours after weekly intravenous doxorubicin
Measure: Count of Participants; unit: Participants
Arm/Group | Dexamethasone + Ondansetron IV | Dexamethasone + Palonosetron IV
Number analyzed (Participants) | 7 | 34
Participants | 3 | 15

3. Secondary Outcome: Number of Days With Emetic Episodes and Rescue Medicines
Time Frame: Up to 3 months
Measure: Median (Full Range); unit: days
Arm/Group | Dexamethasone + Ondansetron IV | Dexamethasone + Palonosetron IV
Number analyzed (Participants) | 7 | 34
days
  Vomiting during neoadjuvant chemotherapy | 0 [0 to 51] | 0 [0 to 51]
  Took rescue medicines | 2 [0 to 70] | 9.5 [0 to 70]

4. Secondary Outcome: Number of Participants That Had Emesis Within 48 Hours of Chemotherapy
Description: Count of patients that had emesis within 48 hours of chemotherapy
Time Frame: Up to 48 hours of chemotherapy
Measure: Count of Participants; unit: Participants
Arm/Group | Dexamethasone + Ondansetron IV | Dexamethasone + Palonosetron IV
Number analyzed (Participants) | 7 | 34
Participants | 0 | 1

5. Secondary Outcome: Number of Participants That Had First Administration of Rescue Medication Within 48 Hours
Description: Count of patients that had first administration of rescue medication within 48 Hours
Time Frame: up to 48 hours of chemotherapy
Measure: Count of Participants; unit: Participants
Arm/Group | Dexamethasone + Ondansetron IV | Dexamethasone + Palonosetron IV
Number analyzed (Participants) | 7 | 34
Participants | 1 | 4

6. Secondary Outcome: Number of Doses of Rescue Medications Used
Time Frame: Days 1-7 of each cycle
Population: Patients were unable to consistently complete this part of the FLIE questionnaire and thus we did not retain data from any of the participants.
Arm/Group | Dexamethasone + Ondansetron IV | Dexamethasone + Palonosetron IV
Number analyzed (Participants) | 0 | 0

7. Secondary Outcome: Side Effects of Antiemetic Medications Used
Time Frame: Up to 3 months
Measure: Count of Participants; unit: Participants
Arm/Group | Dexamethasone + Ondansetron IV | Dexamethasone + Palonosetron IV
Number analyzed (Participants) | 7 | 34
Participants
  Constipation | 2 | 15
  Headaches | 0 | 2

8. Secondary Outcome: Severity of Nausea
Description: Count of participants with severe nausea
Time Frame: Up to 3 months
Measure: Count of Participants; unit: Participants
Arm/Group | Dexamethasone + Ondansetron IV | Dexamethasone + Palonosetron IV
Number analyzed (Participants) | 7 | 34
Participants | 1 | 4

9. Secondary Outcome: Quality of Life
Time Frame: Up to 3 months
Measure: Count of Units; unit: FLIE questionnaires
Units Other Than Participants: FLIE questionnaires
Groups:
- Dexamethasone + Ondansetron IV: Patients receive dexamethasone IV or orally and ondansetron IV on day 1 (prior to each dose of doxorubicin hydrochloride).
- Dexamethasone + Palonosetron IV: Patients receive dexamethasone IV or orally and palonosetron IV on day 1 (prior to each dose of doxorubicin hydrochloride).
Arm/Group | Dexamethasone + Ondansetron IV | Dexamethasone + Palonosetron IV
Number analyzed (Participants) | 7 | 34
Number analyzed (FLIE questionnaires) | 35 | 366
FLIE questionnaires
  FLIE Nausea: High impact (<36) | 4 | 44
  FLIE Nausea: Medium impact (36-54) | 5 | 74
  FLIE Nausea: No impact of daily life (>54) | 26 | 248
  FLIE Vomiting: High impact (<36) | 1 | 10
  FLIE Vomiting: Medium impact (36-54) | 3 | 9
  FLIE Vomiting: No impact of daily life (>54) | 31 | 347

ADVERSE EVENTS:
Arm/Group | Dexamethasone + Ondansetron IV | Dexamethasone + Palonosetron IV
Serious Adverse Events (participants affected / at risk) | 0/7 | 0/34
Other Adverse Events (participants affected / at risk) | 2/7 | 15/34
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Dexamethasone + Ondansetron IV (N=7) | Dexamethasone + Palonosetron IV (N=34)
Constipation (Gastrointestinal disorders) | 2 | 15
Headache (General disorders) | 0 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes